CLINICAL TRIAL: NCT04006834
Title: Hypersomnia in Major Depressive Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Zhang Jihui, Dr., Chinese University of Hong Kong
Other Study IDs: CREC2018.317
Record Dates: First submitted 2019-02-25; First posted 2019-07-05 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MDD with hypersomnia: Patient with a history of MDD and ESS >10
  Interventions: Other: No intervention involved
- MDD without hypersomnia: Patient with a history of MDD and ESS <=10
  Interventions: Other: No intervention involved

INTERVENTIONS:
Other: No intervention involved — No intervention involved

SUMMARY:
Background: MDD is a common mental disorder with significant morbidities and mortalities. Recent local data suggested that depressive disorders have a prevalence of over 12% in females and nearly 7 % in males in Hong Kong general adult population. Other than insomnia, patients with MDD often complained another sleep symptom - hypersomnia (defined as daytime sleepiness or excessive sleep). Interestingly, when compared to insomnia, there is much far less research on the role of hypersomnia in MDD. However, there are available data suggested that hypersomnia is associated with greater treatment-resistance, more recurrence, and increased suicidality, suggesting a need to investigate this problem in MDD patients.

Objective: To investigate the prevalence and determine characteristics of hypersomnia amongst major depressive disorder.

Design: 2-phase study design Setting: A case-control study Participants: Patients with a history of Major Depressive Disorder from out-patient clinics in New Territories East Cluster.

Main outcome measures: Daytime sleepiness measured by MSLT, actigraphy and self-reported questionnaire (ESS), sleep duration as measured by sleep diary and actigraphy.

DETAILED DESCRIPTION:
Background

Significance of hypersomnia in depressive illness

Sleep disturbances are observed in up to 90% of depressed patients. Both insomnia, defined clinically as difficulty initiating and/or maintain sleep, and hypersomnia, defined as excessive daytime sleepiness (EDS) and/or excessive sleep duration, are key symptoms in the diagnostic criteria of depression. A sizeable number of studies have demonstrated clear associations between insomnia and poorer depressive outcomes. These include greater depressive symptom severity, poorer treatment response and increased risk of suicidal ideations and attempts. Persistent insomnia complaints following remission of major depressive episodes (MDE) have also been found to be associated with greater risk of recurrence, poorer overall functioning and quality of life. Compared to insomnia, there is much less research on the role of hypersomnia in depressive illness.

Studies so far have suggested a prognostic significance. Hypersomnia in depressed subjects amongst a mix of mood disorders have been linked to greater treatment-resistance, depressive relapse, higher suicidal ideations and increased risk of suicide; while hypersomnia complaints amongst general populations have predicted the risk of incident depression. More recently, studies of depressed individuals amongst a mix of mood disorders had further found that the concurrence of insomnia and hypersomnia was associated with worse symptomatology compared to patients with insomnia or hypersomnia alone. These studies also found that the concurrence of insomnia and hypersomnia had greater associations with bipolar spectrum features, which builds on from previous findings suggesting that hypersomnia itself may be a clinical marker for undetected or subsequent diagnosis of bipolar II disorders in depressed patients.

Knowledge gaps in the understanding of hypersomnia in major depression

Despite its prognostic implications, there is currently a lack of studies investigating potential determinants or clinical correlates of hypersomnia in major depressive disorder (MDD). MDD is one of the commonest diagnoses encountered in the outpatient setting, and may be distinct in its determinants and outcomes compared to other mood disorders. Existing studies on hypersomnia in depression have predominantly included subjects from a mix of mood disorders; thus, a gap exists to extend the scope of understanding on hypersomnia amongst unipolar depression.

Due to the lack of standardized definitions, even amongst contemporary classifications, there is little clarity as to which aspect of hypersomnia - i.e. whether EDS or excessive sleep duration, or in combination - is related to poorer depressive outcomes. Moreover, little is known about what severity of "excessive" daytime sleepiness and sleep duration may be of clinical significance. Most studies of hypersomnia in mood disorders have used crude definitions, predominantly in form of single yes/no questions, to define hypersomnia. Despite the availability of validated questionnaires such as the Epworth Sleepiness Scale (ESS) that could help quantify EDS, or the use of sleep diaries that may help determine an individual's average sleep duration, limited studies of hypersomnia in MDD have employed these tools. The variability in definitions have also resulted in a large range of reported prevalence - between 8.9% to 78% of hypersomnia in MDD samples. In order to generate more clinically useful data, it may be helpful to "deconstruct" hypersomnia into EDS and prolonged sleep duration, to quantify them using validated or clinically-relevant measures, and further analyze their associations with potential determinants and depressive outcomes.

Theoretically, a myriad of factors can contribute to EDS or prolonged sleep duration. These include physical-health related factors, such as the use of sedative medications, the presence of medical illnesses and sleep-related breathing disorders; also sleep-related factors, such as the need for shift-work, the presence of insomnia or other sleep-behavioral disturbances, or the presence of circadian-disorders or particular chronotype preferences. Psychiatric factors, such as increased anxiety, somatic complaints and perceived fatigue levels, may also be related to EDS or prolonged sleep duration. So far, no studies have simultaneously examined this range of factors and their potential associations with hypersomnia complaints in MDD. Whether these factors mediate or act synergistically with hypersomnia to influence depressive outcomes remain to be elucidated.

A limitation that many hypersomnia studies have faced is the lack of objective measures used to corroborate subjective measures of EDS or sleep duration. The mean sleep latency test (MSLT) is currently regarded as the gold standard objective measure for EDS, while polysomnography (PSG) and wrist actigraphy has been useful in validating sleep diary data. However, the costs, expertise and time required to conduct these tests have limited their use. A study involving the use of both subjective and objective measures of EDS or sleep duration, in addition to a thorough analysis of the potential determinants and clinical correlates, may provide valuable information on the clinical profiles of hypersomnia patients and shed light on areas for further research and management.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18-64 years old with a history of MDD

Exclusion Criteria:

* patients with history of bipolar disorder, schizophrenic-spectrum disorder, substance abuse, alcohol dependence, dementia, patients with history of mental retardation and those unable to give consent.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects will be successively recruited from August 2018 to August 2019 from the out-patient psychiatric clinics within the New Territories Eastern Cluster.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Hypersomnia | 1 year
  Daytime Sleepiness measured by self rated Epworth Sleepiness Scale
Depression severity | 1 year
  Clinician rated score by Structure Interview Guide for the Hamilton Depression Rating Scale - Seasonal Affective Disorder (SIGH-SAD)

SECONDARY OUTCOMES:
Fatigue | 1 year
  Self rated scale by Multidimensional Fatigue Inventory (MFI)
Function as indicated quality of life | 1 year
  Self rated by 12-Item Short FOrm Survey (SF12)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang JiHui, Dr, Principal Investigator — CUHK
Locations (1):
- Department of psychiatry, Faculty of Medicine, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No